CLINICAL TRIAL: NCT06865105
Title: A Phase 2 Multicenter, Randomized, Platform Study of Targeted Therapies for the Treatment of Adult Subjects With Active Psoriatic Arthritis
Brief Title: Study of Targeted Therapies for the Treatment of Adult Participants With Active Psoriatic Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-191
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — lutikizumab; risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sub-Study 1: Risankizumab Monotherapy (Experimental): Participants will receive Risankizumab
  Interventions: Drug: Risankizumab
- Sub-Study 1: Lutikizumab Monotherapy (Experimental): Participants will initially receive Lutikizumab Dose A followed by Lutikizumab Dose B every other week.
  Interventions: Drug: Lutikizumab
- SubStudy 1: Lutikizumab and Risankizumab Combination Therapy (Experimental): Participants will be administered Lutikizumab and Risankizumab at the same time following the same dosing regimen as the monotherapy arms.
  Interventions: Drug: Lutikizumab; Drug: Risankizumab

INTERVENTIONS:
Drug: Lutikizumab — Subcutaneous (SC) Injection
  Arms: Sub-Study 1: Lutikizumab Monotherapy; SubStudy 1: Lutikizumab and Risankizumab Combination Therapy
Drug: Risankizumab — Subcutaneous (SC) Injection
  Arms: Sub-Study 1: Risankizumab Monotherapy; SubStudy 1: Lutikizumab and Risankizumab Combination Therapy

SUMMARY:
Psoriatic arthritis (PsA) is a type of arthritis that happens when the body's immune system attacks healthy cells and tissues causing joint pain, stiffness, and swelling. Symptoms can get worse and go away for periods of time. This study will evaluate the efficacy and safety of targeted therapies through a series of substudies, for the treatment of active psoriatic arthritis and to assess the changes in disease symptoms.

The therapies being assessed in this sub-study are risankizumab and lutikizumab. Participants will be randomized in a 1:1:1 ratio to one of the three treatment arms: lutikizumab monotherapy, risankizumab monotherapy or a combination therapy of lutikizumab and risankizumab. Around 120 participants will be enrolled in the study at approximately 40 sites worldwide.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to comply with procedures required in the Master Protocol and substudies.
* Participant has a documented clinical diagnosis of PsA with symptom onset at least 6 months prior to the Screening Visit and fulfillment of the Classification Criteria for Psoriatic Arthritis (CASPAR) at Screening Visit.
* Participant has active disease defined as greater than or equal to 3 tender joints (based on 68 joint count) and greater than or equal to 3 swollen joints (based on 66 joint count) at both the Screening Visit and Baseline.
* Participant has active plaque PsO and/or a documented history of plaque PsO.
* Participant must demonstrate intolerance or inadequate response to 1 to 2 targeted therapies (biologic or targeted synthetic disease-modifying antirheumatic drugs) approved for the treatment of PsA

Exclusion Criteria:

* Participants who have had major surgery performed within 12 weeks prior to randomization or plan to have a major surgery during conduct of the study (e.g., aneurysm removal, stomach ligation).
* Participants with the following chronic or active infections: Are infected with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus(HCV) infection, active tuberculosis(TB)
* Active skin disease other than psoriasis (PsO) which could interfere with the assessment of PsO.
* History of fibromyalgia, any arthritis with onset prior to age 17 years, or current diagnosis of inflammatory joint disease other than psoriatic arthritis (PsA) (including but not limited to rheumatoid arthritis, gout, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, systemic lupus erythematosus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response | At Week 16
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Number of Participants With Adverse Events (AEs) | Up to Week 52
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Minimal Disease Activity (MDA) Response | At Week 16
  A participant was classified as achieving MDA if 5 of the following 7 criteria were met:
  * Tender joint count (out of 68 joints) ≤ 1
  * Swollen joint count (out of 66 joints) ≤ 1
  * PASI score ≤ 1 (score ranges from 0 - 72) or percent BSA involved with psoriasis ≤ 3%
  * Participant's assessment of pain ≤ 1.5 (NRS from 0 to 10)
  * Participant's Global Assessment of disease activity ≤ 2 (NRS from 0 to 10)
  * HAQ-DI score ≤ 0.5 (index score ranges from 0 to 3)
  * Leeds Enthesitis Index ≤ 1 (assesses the presence or absence of enthesitis at 3 bilateral sites, with an overall score range from 0 to 6)
Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response | At Week 16
  Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response | At Week 16
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 Response (in the subset of participants with a PsO BSA ≥ 3% at Baseline) | At Week 16
  PASI is a composite score based on the percentage of the body surface area (BSA) affected by psoriasis and the intensity of erythema (reddening), induration (thickening or hardening of the skin), and desquamation (peeling of the skin) of lesions assessed at 4 anatomic sites (head, upper extremities, trunk, and lower extremities). At each location, the percentage of BSA involvement is assigned a score from 0 (no involvement) to 6 (90% to 100% involvement), and erythema, induration, and desquamation are scored on a scale from 0 (no symptoms) to 4 (very marked).
  The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from Baseline in PASI score, and was assessed in participants with Baseline psoriasis BSA involvement ≥ 3%.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (16):
  - Newport Huntington Medical Group /ID# 272764, Huntington Beach, California
  - Highlands Advanced Rheumatology And Arthritis Center - Avon Park /ID# 273085, Avon Park, Florida
  - Clinical Research Of West Florida - Phase I Unit /ID# 273198, Clearwater, Florida
  - HMD Research LLC /ID# 273086, Orlando, Florida
  - West Broward Rheumatology Associates /ID# 272892, Tamarac, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 273199, Tampa, Florida
  - Clinic Of Dr. Robert Hozman/Clinical Investigation Specialists, Inc /ID# 272879, Skokie, Illinois
  - Willow Rheumatology and Wellness, PLLC /ID# 277354, Willowbrook, Illinois
  - Klein And Associates /ID# 272829, Hagerstown, Maryland
  - Paramount Medical Research and Consulting /ID# 272757, Middleburg Heights, Ohio
  - Altoona Center For Clinical Research /ID# 272593, Duncansville, Pennsylvania
  - Private Practice - Dr. Ramesh C. Gupta I /ID# 272897, Memphis, Tennessee
  - Tekton Research - West Gate /ID# 272765, Austin, Texas
  - Accurate Clinical Research - Houston /ID# 272754, Houston, Texas
  - Tekton Research, LLC /ID# 272901, San Antonio, Texas
  - Dynamed Clinical Research - Tomball /ID# 272760, Tomball, Texas
- Canada (2):
  - Centre de Recherche Musculo-Squelettique /ID# 274397, Trois-Rivières, Quebec
  - Dr. Latha Naik Medical Professional Corporation /ID# 272803, Saskatoon, Saskatchewan
- Czechia (4):
  - Revmatologie /ID# 272367, Brno, Brno-mesto
  - L.K.N. Arthrocentrum /ID# 272366, Hlučín, Moravskoslezský kraj
  - Medical Plus s.r.o. /ID# 272363, Uherské Hradiště
  - PV Medical Services s.r.o. /ID# 272368, Zlín
- France (5):
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur /ID# 272771, Nice, Alpes-Maritimes
  - Infirmerie Protestante De Lyon /ID# 273731, Caluire-et-Cuire, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional Universitaire De Tours - Hôpital Trousseau /ID# 272762, Chambray-lès-Tours, Indre-et-Loire
  - CHU Bordeaux - Hopital Pellegrin /ID# 273390, Bordeaux, Nouvelle-Aquitaine
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 272877, Orléans
- Hungary (5):
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz /ID# 272572, Miskolc, Borsod-Abauj Zemplen county
  - Complex Rendelo Med Zrt. /ID# 272570, Székesfehérvár, Fejér
  - Vital-Medicina Kft. /ID# 272855, Veszprém, Fejér
  - Semmelweis Egyetem Reumatológiai és Immunológiai Klinika /ID# 273195, Budapest
  - Revita Reumatologiai Rendelo (Revita Kft.) /ID# 272857, Budapest
- Poland (5):
  - Mics Centrum Medyczne Bydgoszcz /ID# 273297, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MCBK S.C. Iwona Czajkowska Anna Podrazka-Szczepaniak /ID# 273305, Pruszków, Masovian Voivodeship
  - Centrum Medyczne Reuma Park /ID# 273301, Warsaw, Masovian Voivodeship
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik /ID# 273304, Bialystok, Podlaskie Voivodeship
  - Centrum Kliniczno-Badawcze J.Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka /ID# 273306, Elblag, Warmian-Masurian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-191